CLINICAL TRIAL: NCT00177697
Title: A Mentor-Based Approach to Long-Term Weight Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01DK058002 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Weight Loss; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

INTERVENTIONS:
Behavioral: behavioral weight loss program

SUMMARY:
The purpose of this study to examine the effect of having a weight loss mentor on long-term weight loss in overweight adults.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 21-55 years of age
3. BMI = 25-35 kg/m2
4. Ability to provide informed consent.
5. Ability to provide consent from their personal physician to participate in this study.

Exclusion Criteria:

1. Reporting regular exercise participation of at least 20 minutes per day on at least 3 days per week during the previous six months. (This study is designed to recruit relatively sedentary adults.)
2. Diabetes, hypothyroidism, or other medical conditions which would affect energy metabolism.
3. Currently pregnant, pregnant within the previous six months, or planning on becoming pregnant within the next 12 months. (Pregnancy will be based on self-report and will be included on the detailed medical history that is completed by subjects.)
4. Non-medicated resting systolic blood pressure >160 mmHg or non-medicated resting diastolic blood pressure >100 mmHg, or taking medication that would affect blood pressure.
5. Taking medication that would affect resting heart rate or the heart rate response during exercise (e.g., beta blockade).
6. Arrhythmia on resting or exercise electrocardiogram that would indicate that vigorous exercise was contraindicated.
7. History of myocardial infarction or valvular disease.
8. History of orthopedic complications that would prevent optimal participation in the exercise component (e.g., heel spurs, severe arthritis).

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174
Dates: Start 1999-09; Study Completion 2002-07

PRIMARY OUTCOMES:
weight loss

SECONDARY OUTCOMES:
fitness
dietary intake
mediators

CONTACTS AND LOCATIONS:
Overall Officials: John M Jakicic, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States